CLINICAL TRIAL: NCT02759120
Title: Study of Clinical Efficacy of Antimicrobial Therapy Strategy Using Pragmatic Design in Idiopathic Pulmonary Fibrosis
Brief Title: CleanUP IPF for the Pulmonary Trials Cooperative
Acronym: CleanUp-IPF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for futility after review of first planned interim analysis.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Duke Clinical Research Institute (Other); University of Chicago (Other); University of Washington (Other); University of Pittsburgh (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504016087; U01HL128954 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; pulmonary fibrosis; antimicrobial therapy; doxycycline; co-trimoxazole
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antimicrobial therapy (Experimental): Co-trimoxazole OR doxycycline
  Interventions: Drug: Antimicrobial therapy: Co-trimoxazole or Doxycycline
- Standard of care (Other): Standard of care for patients with IPF for comparison
  Interventions: Other: No Intervention: Standard of Care

INTERVENTIONS:
Drug: Antimicrobial therapy: Co-trimoxazole or Doxycycline — 160mg trimethoprim/800mg sulfamethoxazole (double strength co-trimoxazole) twice daily plus folic acid 5 mg daily OR doxycycline 100mg once daily if weight < 50 kilograms or 100mg twice daily if weight > 50 kilograms for up to 36 months
  Arms: Antimicrobial therapy
Other: No Intervention: Standard of Care — Standard of care
  Arms: Standard of care

SUMMARY:
The purpose of this study is to compare the effect of standard care, versus standard of care plus antimicrobial therapy (co-trimoxazole or doxycycline), on clinical outcomes in patients diagnosed with idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
This is a randomized, un-blinded, phase III, multi-center clinical trial of an antimicrobial therapy strategy in idiopathic pulmonary fibrosis patients. Our overall hypothesis is that reducing harmful microbial impact with antimicrobial therapy will reduce the risk of non-elective, respiratory hospitalization or death in patients with Idiopathic Pulmonary Fibrosis (IPF).

Subjects will be randomized 1:1 to either receive a prescription drug voucher for oral antimicrobial therapy in the form of one double strength 160 milligrams (mg) trimethoprim/800mg sulfamethoxazole (double strength co-trimoxazole) twice daily plus folic acid 5 mg daily OR doxycycline 100mg once daily if weight < 50 kilograms (kg) or 100mg twice daily if weight > 50 kg. Patients randomized to receive antimicrobial therapy will be given co-trimoxazole unless they have an allergy, contraindication to co-trimoxazole, renal insufficiency (glomerular filtration rate (GFR) < 30 milliliters (ml)), are hyperkalemic (potassium > 5 milliequivalents(mEq)/liter(L)), or are concomitantly taking an angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), or potassium sparing diuretic in which case they will receive doxycycline.

Participation in this study will be between 12 months and 36 months depending on time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 40 years of age
2. Diagnosed with idiopathic pulmonary fibrosis (IPF) by enrolling investigator
3. Signed informed consent

Exclusion Criteria:

1. Received antimicrobial therapy in the past 30 days
2. Contraindicated for antibiotic therapy, including but not exclusive to:

   1. Allergy or intolerance to both tetracyclines AND trimethoprim, sulfonamides or their combination
   2. Allergy or intolerance to tetracyclines AND known potassium level > 5 mEq/L in the past 90 days.

      * If the enrolling physician feels the potassium level has normalized, documentation to that effect must be provided.
   3. Allergy or intolerance to tetracyclines AND concomitant use of angiotensin converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), potassium sparing diuretic, dofetilide, methotrexate, azathioprine, mycophenolate mofetil, cyclophosphamide
   4. Allergy or intolerance to tetracyclines AND known glucose-6-phosphate dehydrogenase deficiency
   5. Allergy or intolerance to tetracyclines AND untreated folate or B12 deficiency
   6. Allergy or intolerance to tetracyclines AND known renal insufficiency (defined as a glomerular filtration rate (GFR) < 30 ml within the previous 90 days)

      * If the enrolling physician feels the renal dysfunction has resolved, documentation to that effect must be provided.
3. Pregnant or anticipate becoming pregnant
4. Use of an investigational study agent for IPF therapy within the past 30 days, or an IV infusion with a half-life of four (4) weeks.
5. Concomitant immunosuppression with azathioprine, mycophenolate, cyclophosphamide, or cyclosporine.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Martinez, MD, MS, Principal Investigator — Weill Cornell Medical Medicine
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - Stanford, Stanford, California
  - Loyola University Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Mayo Clinic, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State, Columbus, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - University of Texas at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - INOVA, Falls Church, Virginia
  - Washington University, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be uploaded in a de-identified manner into BioLINCC with open access for interested investigators
Supporting Information: Study Protocol, SAP
Time Frame: Within a year of the primary paper publication and then indefinitely maintained by BioLINCC
Access Criteria: The data will be open access for interested investigators
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Kim JS, Murray S, Yow E, Anstrom KJ, Kim HJ, Flaherty KR, Martinez FJ, Noth I. Comparison of Pirfenidone and Nintedanib: Post Hoc Analysis of the CleanUP-IPF Study. Chest. 2024 May;165(5):1163-1173. doi: 10.1016/j.chest.2023.11.035. Epub 2023 Nov 27. PMID 38030064
- [Derived] Martinez FJ, Yow E, Flaherty KR, Snyder LD, Durheim MT, Wisniewski SR, Sciurba FC, Raghu G, Brooks MM, Kim DY, Dilling DF, Criner GJ, Kim H, Belloli EA, Nambiar AM, Scholand MB, Anstrom KJ, Noth I; CleanUP-IPF Investigators of the Pulmonary Trials Cooperative. Effect of Antimicrobial Therapy on Respiratory Hospitalization or Death in Adults With Idiopathic Pulmonary Fibrosis: The CleanUP-IPF Randomized Clinical Trial. JAMA. 2021 May 11;325(18):1841-1851. doi: 10.1001/jama.2021.4956. PMID 33974018
- [Derived] Anstrom KJ, Noth I, Flaherty KR, Edwards RH, Albright J, Baucom A, Brooks M, Clark AB, Clausen ES, Durheim MT, Kim DY, Kirchner J, Oldham JM, Snyder LD, Wilson AM, Wisniewski SR, Yow E, Martinez FJ; CleanUP-IPF Study Team. Design and rationale of a multi-center, pragmatic, open-label randomized trial of antimicrobial therapy - the study of clinical efficacy of antimicrobial therapy strategy using pragmatic design in Idiopathic Pulmonary Fibrosis (CleanUP-IPF) clinical trial. Respir Res. 2020 Mar 12;21(1):68. doi: 10.1186/s12931-020-1326-1. PMID 32164673

RESULTS

PARTICIPANT FLOW:
Groups:
- Antimicrobial Therapy Plus Standard of Care: Co-trimoxazole OR doxycycline
  Antimicrobial therapy: Co-trimoxazole or Doxycycline: 160mg trimethoprim/800mg sulfamethoxazole (double strength co-trimoxazole) twice daily plus folic acid 5 mg daily OR doxycycline 100mg once daily if weight < 50 kilograms or 100mg twice daily if weight > 50 kilograms for up to 36 months
Period: Overall Study
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Started | 254 | 259
Completed | 169 | 180
Not Completed | 85 | 79
Not completed — Death | 34 | 36
Not completed — Lost to Follow-up | 4 | 7
Not completed — Physician Decision | 3 | 0
Not completed — Withdrawal by Subject | 28 | 15
Not completed — Moved out of area | 3 | 4
Not completed — Lung transplant | 3 | 5
Not completed — Other reason not completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 254 | 259 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 92
  >=65 years | 206 | 215 | 421
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 51 | 111
  Male | 194 | 208 | 402
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 241 | 249 | 490
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 231 | 244 | 475
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 254 | 259 | 513
Medical History [Count of Participants; unit: Participants] — Population: Data could not be located.
  Participants
    Coronary artery disease | 69 | 79 | 148
    Myocardial infarct: number analyzed (Participants) | 251 | 259 | 510
    Myocardial infarct | 20 | 32 | 52
    Valvular heart disease: number analyzed (Participants) | 252 | 256 | 508
    Valvular heart disease | 7 | 13 | 20
    Congestive heart failure: number analyzed (Participants) | 254 | 258 | 512
    Congestive heart failure | 8 | 12 | 20
    Stroke: number analyzed (Participants) | 254 | 258 | 512
    Stroke | 9 | 10 | 19
    Osteoarthritis: number analyzed (Participants) | 251 | 256 | 507
    Osteoarthritis | 66 | 73 | 139
    Osteoporosis: number analyzed (Participants) | 252 | 258 | 510
    Osteoporosis | 19 | 11 | 30
    Hypertension: number analyzed (Participants) | 252 | 258 | 510
    Hypertension | 127 | 129 | 256
    High cholesterol: number analyzed (Participants) | 252 | 257 | 509
    High cholesterol | 144 | 154 | 298
    Stomach ulcers: number analyzed (Participants) | 253 | 257 | 510
    Stomach ulcers | 12 | 16 | 28
    Hay fever: number analyzed (Participants) | 250 | 253 | 503
    Hay fever | 51 | 46 | 97
    Atrial fibrillation: number analyzed (Participants) | 252 | 258 | 510
    Atrial fibrillation | 21 | 31 | 52
    Intermittent claudication: number analyzed (Participants) | 248 | 258 | 506
    Intermittent claudication | 2 | 7 | 9
    Peripheral vascular disease: number analyzed (Participants) | 247 | 259 | 506
    Peripheral vascular disease | 9 | 11 | 20
    Cerebrovascular disease: number analyzed (Participants) | 252 | 259 | 511
    Cerebrovascular disease | 3 | 4 | 7
    Dementia | 0 | 3 | 3
    Chronic pulmonary disease | 151 | 163 | 314
    Connective tissue disease: number analyzed (Participants) | 249 | 258 | 507
    Connective tissue disease | 2 | 1 | 3
    Ulcer disease: number analyzed (Participants) | 253 | 257 | 510
    Ulcer disease | 4 | 3 | 7
    Mild liver disease: number analyzed (Participants) | 253 | 258 | 511
    Mild liver disease | 7 | 5 | 12
    Diabetes | 49 | 39 | 88
    Hemiplegia: number analyzed (Participants) | 252 | 258 | 510
    Hemiplegia | 0 | 1 | 1
    Moderate or sever renal disease: number analyzed (Participants) | 253 | 259 | 512
    Moderate or sever renal disease | 9 | 8 | 17
    Diabetes with end organ damage: number analyzed (Participants) | 253 | 259 | 512
    Diabetes with end organ damage | 0 | 1 | 1
    Any tumor | 21 | 16 | 37
    Leukemia | 0 | 1 | 1
    Moderate or severe disease: number analyzed (Participants) | 253 | 258 | 511
    Moderate or severe disease | 4 | 3 | 7
    Metastatic solid tumor | 1 | 0 | 1
    AIDS | 0 | 0 | 0
    Lung cancer | 3 | 4 | 7
    Other cancer (excluding basal cell carcinoma) | 39 | 37 | 76
    Gastroesophageal reflux disease (GERD): number analyzed (Participants) | 251 | 256 | 507
    Gastroesophageal reflux disease (GERD) | 156 | 149 | 305
    Asthma: number analyzed (Participants) | 253 | 257 | 510
    Asthma | 14 | 12 | 26
    Evidence of pulmonary hypertension: number analyzed (Participants) | 253 | 254 | 507
    Evidence of pulmonary hypertension | 19 | 21 | 40
    Emphysema or chronic bronchitis | 25 | 28 | 53
    Lymphoma: number analyzed (Participants) | 253 | 259 | 512
    Lymphoma | 1 | 2 | 3
Physical Exam [Count of Participants; unit: Participants] — Population: Data could not be located.
  Participants
    Clubbing: number analyzed (Participants) | 253 | 256 | 509
    Clubbing | 41 | 51 | 92
    Bibasilar, inspiratory crackles: number analyzed (Participants) | 252 | 259 | 511
    Bibasilar, inspiratory crackles | 238 | 240 | 478
    Jugular venous distension | 4 | 4 | 8
    Increased P2: number analyzed (Participants) | 240 | 251 | 491
    Increased P2 | 7 | 8 | 15
    Peripheral edema | 16 | 20 | 36
    Other significant finding | 13 | 10 | 23
Standard of Care medications [Count of Participants; unit: Participants] — Population: Data could not be located.
  Participants
    Pirfenidone: number analyzed (Participants) | 253 | 259 | 512
    Pirfenidone | 158 | 160 | 318
    Nintedanib: number analyzed (Participants) | 253 | 259 | 512
    Nintedanib | 101 | 97 | 198
Prior medications [Count of Participants; unit: Participants] — Population: Data could not be located.
  Participants
    Proton pump inhibitors (PPI): number analyzed (Participants) | 253 | 259 | 512
    Proton pump inhibitors (PPI) | 158 | 158 | 316
    H2 blockers (H2 receptor antagonists): number analyzed (Participants) | 253 | 259 | 512
    H2 blockers (H2 receptor antagonists) | 49 | 53 | 102
    Chronic prednisone (> 1 month): number analyzed (Participants) | 253 | 259 | 512
    Chronic prednisone (> 1 month) | 43 | 53 | 96
    Azathioprine: number analyzed (Participants) | 253 | 259 | 512
    Azathioprine | 1 | 3 | 4
    N-acetylcysteine (NAC): number analyzed (Participants) | 253 | 259 | 512
    N-acetylcysteine (NAC) | 14 | 13 | 27
    Co-trimoxazole: number analyzed (Participants) | 253 | 259 | 512
    Co-trimoxazole | 43 | 38 | 81
    Doxycycline: number analyzed (Participants) | 253 | 259 | 512
    Doxycycline | 54 | 41 | 95
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Liters] — Population: Data could not be located.
  Liters
    number analyzed (Participants) | 247 | 255 | 502
    (all) | 2.20 (0.621) | 2.23 (0.624) | 2.22 (0.622)
Forced expiratory volume in 1 second (FEV1) percent predicted [Mean (Standard Deviation); unit: percent predicted] — Population: Data could not be located.
  percent predicted
    number analyzed (Participants) | 237 | 254 | 491
    (all) | 78.79 (19.656) | 77.01 (18.195) | 77.87 (18.916)
Forced expiratory volume (FEV1)/Forced vital capacity (FVC) percentage [Mean (Standard Deviation); unit: percent] — Population: Data could not be located.
  percent
    number analyzed (Participants) | 242 | 258 | 500
    (all) | 73.68 (2.138) | 73.46 (2.098) | 73.57 (2.118)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: Liters] — Population: Data could not be located.
  Liters
    number analyzed (Participants) | 247 | 255 | 502
    (all) | 2.71 (0.798) | 2.78 (0.848) | 2.75 (0.824)
Forced vital capacity (FVC) percent predicted [Mean (Standard Deviation); unit: percent predicted] — Population: Data could not be located.
  percent predicted
    number analyzed (Participants) | 237 | 254 | 491
    (all) | 71.36 (18.071) | 70.20 (17.683) | 70.76 (17.863)
Diffusing capacity of the lung for carbon monoxide (DCLO) [Mean (Standard Deviation); unit: mL/min/mmHg] — Population: Data could not be located.
  mL/min/mmHg
    number analyzed (Participants) | 240 | 252 | 492
    (all) | 11.50 (4.630) | 11.74 (4.414) | 11.62 (4.518)
Diffusing capacity of the lung for carbon monoxide (DLCO) corrected [Mean (Standard Deviation); unit: mL/min/mmHg] — Population: Data could not be located.
  mL/min/mmHg
    number analyzed (Participants) | 185 | 192 | 377
    (all) | 11.42 (4.323) | 192 (4.466) | 11.59 (4.393)
Diffusing capacity of the lung for carbon monoxide (DLCO) percent predicted (actual) [Mean (Standard Deviation); unit: percent predicted] — Population: Data could not be located.
  percent predicted
    number analyzed (Participants) | 233 | 251 | 484
    (all) | 40.48 (16.738) | 39.78 (13.832) | 40.11 (15.288)
Diffusing capacity of the lung for carbon monoxide (DLCO) percent predicted (corrected) [Mean (Standard Deviation); unit: percent] — Population: Data could not be located.
  percent
    number analyzed (Participants) | 179 | 191 | 370
    (all) | 40.20 (15.040) | 40.00 (13.988) | 40.10 (14.487)
Diffusing capacity of the lung for carbon monoxide (DLCO) percent predicted (best available) [Mean (Standard Deviation); unit: percent] — Population: Data could not be located.
  percent
    number analyzed (Participants) | 233 | 251 | 484
    (all) | 40.68 (16.939) | 40.11 (13.814) | 40.38 (15.384)
GAP stage [Number; unit: participants] — The GAP stage assessment system is a clinical prediction tool that estimates prognosis in patients with idiopathic pulmonary fibrosis. The GAP model includes four baseline variables that were found to be predictive of outcome, as identified by logistic regression. These factors are: gender (G), age (A) and two lung physiology variables (P) (forced vital capacity and diffusing capacity of the lung for carbon monoxide). A higher stage indicates a higher rate of mortality.
  One year mortality rates by stage:
  Stage I = 6% Stage II=16% Stage III = 39% Population: Data could not be located.
  participants
    I: number analyzed (Participants) | 233 | 251 | 484
    I | 60 | 54 | 144
    II: number analyzed (Participants) | 233 | 251 | 484
    II | 124 | 133 | 257
    III: number analyzed (Participants) | 233 | 251 | 484
    III | 49 | 64 | 113
University of California San Diego (UCSD) shortness of breath questionnaire total score [Mean (Standard Deviation); unit: Scores on a scale] — University of California San Diego (UCSD) Shortness of Breath Questionnaire (SOBQ) total score (0 - 120 range). A lower score indicates a better health score.
  The UCSD SOBQ is a 24-item self-administered questionnaire that assesses dyspnea associated with activities of daily living. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 251 | 257 | 508
    (all) | 32.62 (24.246) | 32.91 (32.91) | 32.77 (32.77)
EuroQoL index score [Mean (Standard Deviation); unit: Scores on a scale] — EuroQoL score (0 - 1 range). A higher score indicates a better health score.
  This self-administered instrument includes five health state items (e.g. mobility, self-care). Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 250 | 255 | 505
    (all) | 0.80 (0.191) | 0.80 (0.173) | 0.80 (0.182)
EuroQoL thermometer response [Mean (Standard Deviation); unit: Scores on a scale] — EuroQoL visual analog scale (0 - 100 range). A higher score indicates a better health score.
  Includes a 0-100 "thermometer" rating of current state of health from 0 as worst imaginable to 100 as best. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 218 | 212 | 430
    (all) | 68.90 (22.286) | 69.78 (20.044) | 69.33 (21.190)
ICEpop CAPability Measure for Older People (ICECAP-O) Score summary score [Mean (Standard Deviation); unit: Scores on a scale] — ICEpop CAPability Measure for Older People (ICECAP-O) Score (0 - 1 range). A lower score indicates a better health score. The ICECAP-O is a measure of capability in older people for use in economic evaluation. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 253 | 258 | 511
    (all) | 0.35 (0.217) | 0.36 (0.209) | 0.36 (0.213)
SF12 mental component summary (MCS) score [Mean (Standard Deviation); unit: score on a scale] — Short Form-12 mental component summary (MCS) score (0 - 100 range). A higher score indicates a better health score.
  The Short Form 12 MSC score assess mental health and well-being. Population: Data could not be located.
  score on a scale
    number analyzed (Participants) | 252 | 258 | 510
    (all) | 0.35 (0.217) | 0.36 (0.209) | 0.36 (0.213)
SF12 physical component summary (PCS) score [Mean (Standard Deviation); unit: Scores on a scale] — Short form-12 physical components summary (PSC) score (0 - 100 range). A higher score indicates a better health score.
  The Short form-12 PSC score assesses limitations in physical activity because of health problems. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 251 | 258 | 509
    (all) | 41.46 (8.776) | 40.23 (9.171) | 40.83 (8.991)
SF6D score (economic evaluation) [Mean (Standard Deviation); unit: Scores on a scale] — Short form-12 6D health survey score (0.29 - 1.00 range). A higher score indicates a better health score.
  The Short form-12 6D health survey provides an economical evaluation. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 249 | 258 | 507
    (all) | 0.72 (0.115) | 0.72 (0.114) | 0.72 (0.115)
Fatigue Severity Scale score [Mean (Standard Deviation); unit: Scores on a scale] — Fatigue Severity Score (1 - 7 range). A lower score indicates a better health score. The fatigue severity questionnaire measures how fatigue impacts one's ability to function in the last week. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 252 | 253 | 505
    (all) | 3.81 (1.554) | 3.98 (1.708) | 3.90 (1.633)
Leicester cough questionnaire total score [Mean (Standard Deviation); unit: Scores on a scale] — Leicester cough questionnaire total score (3 - 21 range). A higher score indicates a better health score.
  The Leicester cough questionnaire assesses symptoms of cough frequency and severity. Population: Data could not be located.
  Scores on a scale
    number analyzed (Participants) | 249 | 257 | 506
    (all) | 16.71 (3.681) | 17.19 (3.589) | 16.95 (3.638)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Non-elective, Respiratory Hospitalization or All-cause Mortality
Time Frame: Randomization to up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Participants | 52 | 56
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.83, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.71 to 1.53]

2. Secondary Outcome: Number of Participants With Death From Any Cause
Time Frame: Randomization to up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Participants | 37 | 37
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.65, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.70 to 1.78]

3. Secondary Outcome: Number of Participants With First Non-elective, Respiratory Hospitalization
Time Frame: Randomization to up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Participants | 36 | 31
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.25, Regression, Cox; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.82 to 2.17]

4. Secondary Outcome: Number of Participants With First Non-elective, All-cause Hospitalization
Time Frame: Randomization to up to 35 months
Measure: Count of Participants; unit: Participants
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Participants | 54 | 47
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.13, Regression, Cox; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.91 to 2.01]

5. Secondary Outcome: Total Number of Non-elective Respiratory Hospitalizations
Time Frame: Randomization to up to 35 months
Measure: Number; unit: hospitalizations
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
hospitalizations | 55 | 43
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.40, Regression, Cox; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.78 to 1.89]

6. Secondary Outcome: Total Number of Non-elective All-cause Hospitalizations
Time Frame: Randomization to up to 35 months
Measure: Number; unit: hospitalizations
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
hospitalizations | 72 | 52
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.16, Regression, Cox; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.90 to 1.83]

7. Secondary Outcome: Percent Change in Forced Vital Capacity (FVC)
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
percent change | -2.99 [-4.23 to -1.75] | -4.13 [-5.28 to -2.98]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.19, Regression, Cox; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-0.56 to 2.83]

8. Secondary Outcome: Percent Change in Diffusion Capacity of Lungs for Carbon Monoxide (DLCO)
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
percent change | -1.72 [-3.27 to -0.18] | -2.56 [-4.54 to -0.59]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.51, Regression, Cox; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-1.67 to 3.35]

9. Secondary Outcome: Total Number of Respiratory Infections
Time Frame: Randomization to up to 35 months
Measure: Number; unit: respiratory infections
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
respiratory infections | 34 | 49
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.13, Regression, Cox; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.46 to 1.11]

10. Secondary Outcome: Change in UCSD-Shortness of Breath Questionnaire
Description: Change in University of California San Diego (UCSD) Shortness of Breath Questionnaire (0 - 120 range). A lower score indicates a better health score. The UCSD-Shortness of Breath Questionnaire assesses the severity of shortness of breath during specific activities of daily living.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | 5.67 [2.75 to 8.59] | 6.29 [3.54 to 9.04]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.76, Regression, Cox; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-4.64 to 3.39]

11. Secondary Outcome: Change in Fatigue Severity Scale Score
Description: Fatigue Severity Scale score (1 - 7 range). A lower score indicates a better health score. The Fatigue Severity Scale measures the severity of fatigue and its effect on a person's activities and lifestyle.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | 0.24 [-0.02 to 0.49] | 0.13 [-0.12 to 0.37]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.54, Regression, Cox; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.24 to 0.46]

12. Secondary Outcome: Change in Leicester Cough Questionnaire Score
Description: Leicester Cough Questionnaire score (3 - 21 range). A higher score indicates a better health score. The Leicester Cough Questionnaire measures quality of life in people with a chronic cough.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | -0.58 [-1.15 to 0.00] | -0.58 [-1.13 to -0.04]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.99, Regression, Linear; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.79 to 0.80]

13. Secondary Outcome: Change in EuroQol Index (EQ-5D) Score
Description: European Quality of Life-5 dimensions (EQ-5D) score (0 - 1 range). A higher score indicates a better health score. The EQ-5D measures quality of life across 5 dimensions (1. Mobility, 2. Self-care, 3. Usual activities, 4. Pain/discomfort, 5. Anxiety/depression.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | -0.040 [-0.071 to -0.009] | -0.046 [-0.075 to -0.016]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.76, Regression, Cox; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-4.64 to 3.39]

14. Secondary Outcome: Change in ICEpop CAPability Measure for Older People (ICECAP-O) Score
Description: Change in ICEpop (Investigating Choice Experiments for the Preferences of Older People) CAPability measure for Older people (ICECAP-O) score (0 - 1 range). A lower score indicates a better health score. The ICEpop CAPability measure for Older people (ICECAP-O) is intended for use in economic evaluations of care services for older people.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | 0.027 [-0.003 to 0.057] | 0.017 [-0.011 to 0.045]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.63, Regression, Cox; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.031 to 0.051]

15. Secondary Outcome: Change in Short Form-12 Health Survey (SF-12) 6D Score
Description: Change in Short Form-12 health survey (SF-12) 6D score (0.29 - 1.00 range). A higher indicates a better health score. The SF-12 6D score provides and economic evaluation.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | -0.013 [-0.031 to 0.005] | -0.031 [-0.048 to -0.014]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.15, Regression, Cox; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.007 to 0.043]

16. Secondary Outcome: Change in Short Form-12 Health Survey (SF-12) Physical Score
Description: Change in short form-12 health survey (SF-12) physical component summary (PSC) score (0 - 100 range). A higher score indicates a better health score.
  The short form-12 health survey physical score assesses limitations in physical activities because of health problems.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | -1.36 [-2.54 to -0.18] | -1.88 [-3.00 to -0.75]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.53, Regression, Cox; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-1.11 to 2.15]

17. Secondary Outcome: Change in SF-12 Health Survey (SF-12) Mental Score
Description: Change in short form-12 health survey (SF-12) mental component summary (MCS) score (0 - 100 range). A higher score indicates a better health score.
  The short form-12 health survey (SF-12) mental component summary (MCS) assesses general mental health.
Time Frame: Randomization to 12 months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
Number analyzed (Participants) | 254 | 259
Scores on a scale | -1.29 [-2.67 to 0.09] | -1.59 [-2.91 to -0.27]
Statistical Analysis 1: Comparison: Standard of Care; Test type: Superiority; p = 0.75, Regression, Linear; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.61 to 2.20]

ADVERSE EVENTS:
Time Frame: Thirty-five months
Arm/Group | Antimicrobial Therapy Plus Standard of Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 37/254 | 37/259
Serious Adverse Events (participants affected / at risk) | 71/254 | 65/259
Other Adverse Events (participants affected / at risk) | 62/254 | 23/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antimicrobial Therapy Plus Standard of Care (N=254) | Standard of Care (N=259)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 5 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary embollism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 5 (5) | 7 (7)
Cardiac disorder (Cardiac disorders) | 11 (12) | 11 (11)
Nervous system disorder (Nervous system disorders) | 8 (8) | 3 (3)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 42 (51) | 26 (29)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 4 (4)
General disorders and administrative site conditions (General disorders) | 5 (6) | 1 (1)
Metabolic and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Vascular disorders (Vascular disorders) | 3 (3) | 1 (1)
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 0 (0)
Neoplasm benign, malignant, and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0)
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1)
Investigations (Investigations) | 0 (0) | 1 (2)
Product issues (Product Issues) | 0 (0) | 1 (1)
Infections and infestations (Infections and infestations) | 7 (9) | 17 (17)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antimicrobial Therapy Plus Standard of Care (N=254) | Standard of Care (N=259)
Arrhythmia (Cardiac disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (14) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (11) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 17 (22) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 26 (29) | 8 (8)
Other (General disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02759120/SAP_000.pdf
  • Study Protocol (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT02759120/Prot_001.pdf